CLINICAL TRIAL: NCT07333625
Title: Integrating Spiritual Care Into Type 2 Diabetes Management: Effects on Psychological Resilience, Distress, and Glycemic Control
Brief Title: Spiritual Care for Psychological and Glycemic Outcomes in Type 2 Diabetes
Acronym: SC-DMT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Noor Huda Mustofa (Other)
Responsible Party: Principal Investigator, Faisal Amir, Universitas Noor Huda Mustofa, Universitas Noor Huda Mustofa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC-DMT2-2024-AMM; 1853/KEPK/STIKES-NHM/EC/V/2023 (Other: STIKES Ngudia Husada Madura)
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spiritual Care Plus Standard Care (Experimental): Participants received standard diabetes care combined with a structured spiritual care program.
  Interventions: Behavioral: Spiritual Care Program; Behavioral: Standard Diabetes Care
- Standard Diabetes Care (Active Comparator): Participants received standard diabetes care without additional spiritual care intervention.
  Interventions: Behavioral: Standard Diabetes Care

INTERVENTIONS:
Behavioral: Spiritual Care Program — A structured spiritual care program integrated into standard diabetes management, including guided spiritual reflection, supportive counseling, and meaning-centered support delivered by trained healthcare providers.
  Arms: Spiritual Care Plus Standard Care
Behavioral: Standard Diabetes Care — Standard diabetes management provided according to hospital clinical guidelines, including medical treatment, dietary counseling, and routine diabetes education.

SUMMARY:
This study aims to evaluate the effects of integrating spiritual care into the management of patients with type 2 diabetes mellitus. The study examines whether a structured spiritual care program can improve psychological resilience, reduce psychological distress, and help control blood glucose levels in adults with type 2 diabetes. Participants receive standard diabetes care, with one group also receiving spiritual care interventions delivered by trained health professionals. The findings of this study are expected to support a more holistic approach to diabetes management that addresses both physical and psychological well-being.

DETAILED DESCRIPTION:
This study is a randomized controlled clinical trial designed to evaluate the impact of integrating spiritual care into standard management for adults with type 2 diabetes mellitus. Psychological distress and reduced resilience are common among patients with chronic illnesses such as diabetes and may negatively influence glycemic control. Integrating spiritual care into routine diabetes management may help address these psychosocial challenges and improve overall patient well-being.

Eligible participants with type 2 diabetes mellitus were randomly assigned to one of two groups. The experimental group received standard diabetes care combined with a structured spiritual care program, while the control group received standard diabetes care alone. The spiritual care intervention was delivered by trained health professionals and included supportive spiritual counseling, reflective practices, and discussions tailored to patients' beliefs and coping needs.

Primary outcomes of the study included changes in psychological resilience, psychological distress, and glycemic control as measured by blood glucose levels. Secondary outcomes included additional psychological and clinical indicators relevant to diabetes management. Outcome assessments were conducted at baseline and after completion of the intervention period.

The study was conducted in a hospital setting in Indonesia and followed ethical principles for research involving human participants, with approval obtained from an institutional ethics committee. The findings are expected to provide evidence to support holistic and patient-centered approaches to diabetes care that integrate spiritual and psychological dimensions alongside standard medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can read and communicate well;
* Clinically diagnosed with type II di-abetes; and
* Patients over the age of 40
* Willing to participate and provide written informed consent

Exclusion Criteria:

* Diagnosed with severe psychiatric disorders
* Having cognitive impairment that interferes with participation

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-06-02 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Psychological Resilience | Baseline and post-intervention (4 weeks)
  Psychological resilience measured using a validated resilience questionnaire, with higher scores indicating greater resilience.
Psychological Distress | Baseline and post-intervention (4 weeks)
  Psychological distress assessed using a standardized psychological distress scale, with higher scores indicating greater distress.
Blood Glucose Level | Baseline and post-intervention (4 Weeks)
  Fasting blood glucose level measured in milligrams per deciliter (mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Amir, Principal Investigator — Universitas Noor Huda Mustofa
Locations (1):
- RSU Anna Medika Madura, Bangkalan, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koenig HG. Religion, spirituality, and health: the research and clinical implications. ISRN Psychiatry. 2012 Dec 16;2012:278730. doi: 10.5402/2012/278730. Print 2012. PMID 23762764